CLINICAL TRIAL: NCT04106544
Title: A Prospective and Retrospective Cohort Study to Refine and Expand the Knowledge on Patients With Chronic Forms of Acid Sphingomyelinase Deficiency (ASMD)
Brief Title: A Prospective and Retrospective Cohort Study in Patients With Chronic Forms of Acid Sphingomyelinase Deficiency (ASMD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PIR16183
Record Dates: First submitted 2019-09-04; First posted 2019-09-27 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Sphingomyelin Lipidosis
MeSH Terms: conditions — Niemann-Pick Disease, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acid Sphingomyelinase Deficiency (ASMD) Cohort (Other): Patients across the full spectrum of chronic ASMD who have fulfilled the eligibility criteria and who have performed the inclusion visit
  Interventions: Procedure: Investigational Procedures

INTERVENTIONS:
Procedure: Investigational Procedures — The investigational assessments will be performed

SUMMARY:
Primary Objective:

* To describe the clinical features and their severity at the time of diagnosis and their evolution over time in patients with confirmed chronic visceral and chronic neurovisceral forms of ASMD
* To describe Clinician-Reported Outcomes (ClinROs) and Patient-Reported Outcomes (PROs) at enrollment and their evolution over time; disease severity at the time of diagnosis and its evolution over time

Secondary Objectives:

* To describe abnormal values in laboratory parameters and all values of specific clinical and imaging assessments at the time of diagnosis and their evolution over time
* To study the use and applicability towards validation of a newly developed ASMD disease severity scoring system
* To study the use and applicability towards validation of a newly developed ASMD PRO tool
* To describe ASMD-related disease burden among patients with ASMD, caregivers, and healthcare resource utilization
* To describe the association between patient demographics (eg, age, gender, race, Ashkenazi ancestry) and genotype with selected clinical features in patients with confirmed chronic visceral and chronic neurovisceral forms of ASMD

DETAILED DESCRIPTION:
Estimated average of study duration (for each patient) is 2 years

ELIGIBILITY:
Inclusion criteria :

* Patients with confirmed diagnosis of chronic forms of ASMD based on 1) a clinical diagnosis consistent with chronic visceral ASMD (ie, NPD B) or chronic neurovisceral ASMD (ie, NPD B variant or intermediate NPD A/B) and 2) deficient enzymatic activity (as measured in peripheral leukocytes, cultured fibroblasts, lymphocytes, or DBS) or presence of 2 pathogenic SMPD1 mutations,
* The patient (or patient's legal guardian) must provide signed informed consent.

Exclusion criteria:

Patients suspected or diagnosed with infantile onset ASMD (ie, NPD A, with progressive developmental delay, or presence of any combination of R498L, L304P, and P333fs*52 genotypes, if available),

* Patients having received or receiving an investigational drug,
* Patients receiving any ASMD specific ERT,
* Patients with poor general condition that would not be able to undergo study assessments as per investigator's clinical judgment.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2019-09-27 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Time of first occurrence and recurrence of the clinical features and medical interventions related to chronic ASMD | Minimum 2 years
Number of patients with at least one clinical feature and highest severity grade at the time of diagnosis and over time | Minimum 2 years
Clinician-Reported Outcomes (ClinROs) depending on participant's age, local regulation, local availability and investigator's discretion | Up to 2 years
  Clinical Global Impression rating scale (CGI, modified), Neuropathy Symptoms Score (NSS) , Neuropathy Disability Score(NDS), Brief Ataxia Rating Scale (BARS), The Essential Tremor Rating Assessment Scale (TETRAS), Wechsler Preschool and Primary Scale of Intelligence - Fourth Edition (WPPSI™ - IV) , Wechsler Intelligence Scale for Children - Fifth Edition (WISC®-V) and Mini-Mental State Examination (MMSE)
Patient-Reported Outcomes (PROs) depending on participant's age, local regulation, local availability and investigator's discretion | Up to 2 years
  EuroQol-5D-5L , EQ-5D-Y, Pediatric Quality of Life Inventory (PedsQL) core module, 36-Item Short Form Health Survey (SF-36) version 2 , MMRC dyspnea score, PedsQL Multidimensional Fatigue Scale, PedsQL Pediatric Pain Questionnaire, splenomegaly-related symptoms (SRS) v3, Patient Global Impression of Change (PGIC), Patient Global Impression of Symptom Severity (PGIS)

SECONDARY OUTCOMES:
Number of patients with at least one abnormal value in laboratory parameters | Minimum 2 years
Forced vital capacity (FVC) level over time since the time of diagnosis | Minimum 2 years
Forced expiratory volume in the first second of the maneuver (FEV1) | Minimum 2 years
Total lung capacity (TLC) | Minimum 2 years
Diffusion capacity of CO (DLCO) Test | Minimum 2 years
Pulse Oximetry: Saturation of Peripheral Oxygen (SpO2) | Minimum 2 years
Liver volume | Minimum 2 years
Liver stiffness score | Minimum 2 years
Spleen volume | Minimum 2 years
Bone maturation for age (pediatric patients only) | Minimum 2 years
Age appropriate Z-score deviation for height and weight (children only) | Minimum 2 years
Body mass index (BMI) for adults only | Minimum 2 years
Optimization and validation of ASMD disease severity scoring system (DS3) | Up to 2 years
Validation of ASMD PRO instruments (24h and 7-day recall) | UP to 2 years
Niemann-Pick B Health Assessment Questionnaire | UP to 2 years
Health-related Productivity Questionnaire | UP to 2 years
Association of hepatomegaly with age, gender, race, Ashkenazi ancestry and genotype | Minimum 2 years
Association of splenomegaly with age, gender, race, Ashkenazi ancestry and genotype | Minimum 2 years
Association of lower respiratory tract infection with age, gender, race, Ashkenazi ancestry and genotype | Minimum 2 years
Association of respiratory distress with age, gender, race, Ashkenazi ancestry and genotype | Minimum 2 years
Association of oxygen therapy with age, gender, race, Ashkenazi ancestry and genotype | Minimum 2 years
Association of external bleeding episode with age, gender, race, Ashkenazi ancestry and genotype | Minimum 2 years
Association of myocardial infarction with age, gender, race, Ashkenazi ancestry and genotype | Minimum 2 years
Association of cerebrovascular accident with age, gender, race, Ashkenazi ancestry and genotype | Minimum 2 years
Association of hospitalization with age, gender, race, Ashkenazi ancestry and genotype | Minimum 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (28):
- United States (3):
  - Investigational Site Number :8400002, Atlanta, Georgia
  - Investigational Site Number :8400003, The Bronx, New York
  - Investigational Site Number :8400001, Valhalla, New York
- Argentina (2):
  - Investigational Site Number :0320002, CABA
  - Investigational Site Number :0320001, Córdoba
- Investigational Site Number :0560001, Leuven, Belgium
- Brazil (3):
  - Investigational Site Number :0760001, Porto Alegre, Rio Grande do Sul
  - Investigational Site Number :0760002, São Paulo
  - Investigational Site Number :0760006, São Paulo
- Chile (2):
  - Investigational Site Number :152001, Santiago
  - Investigational Site Number :152002, Santiago
- Investigational Site Number :2030001, Prague, Czechia
- France (3):
  - Investigational Site Number :2500002, Angers
  - Investigational Site Number :2500003, Paris
  - Investigational Site Number :2500001, Paris
- Germany (2):
  - Investigational Site Number :2760002, Giessen
  - Investigational Site Number :2760005, Mainz
- Italy (2):
  - Investigational Site Number :380002, Napoli
  - Investigational Site Number :380001, Udine
- Portugal (2):
  - Investigational Site Number :6200001, Porto
  - Investigational Site Number :6200002, Porto
- Investigational Site Number :6420001, Timișoara, Romania
- Spain (3):
  - Investigational Site Number :7240005, Barcelona
  - Investigational Site Number :7240001, Madrid
  - Investigational Site Number :7240004, Seville
- Turkey (Türkiye) (3):
  - Investigational Site Number :7920005, Adana
  - Investigational Site Number :7920003, Istanbul
  - Investigational Site Number :7920001, Izmir

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org